CLINICAL TRIAL: NCT05847881
Title: Toward Thriving: A Set of Reflective Tools to Empower Chronic Pain Patients and Help Them Envision a Personal Path to Thriving.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Center for Advancing Translational Sciences (NCATS) (NIH)
Responsible Party: Principal Investigator, Hannah Smotrich, Associate Professor of Art and Design, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00176302; UM1TR004404 (NIH)
Record Dates: First submitted 2023-04-25; First posted 2023-05-08 (Actual); Results first posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Chronic Pain
Keywords: Positive psychology intervention
MeSH Terms: conditions — Chronic Pain

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Reflective process group (Experimental)
  Interventions: Behavioral: Self-guided at home activities

INTERVENTIONS:
Behavioral: Self-guided at home activities — After the kick-off meeting participants will complete the cultural probe kit for 3 weeks. This kit is a design research tool, to prompt participants to document, map, journal, and reflect on various aspects of daily lives. Following this, participants will attend a facilitated workshop and then complete the next at-home kits.

SUMMARY:
The purpose of this study is to introduce and test the usefulness of a reflective process meant to empower people with chronic pain and help support participant's resiliency and thriving.

The study team hypothesizes that:

-Greater or equal to 80 percent of participants will report that the intervention was relatively easy to understand after orientation, low burden, potentially effective, and will have completed at least 2 of the 3 reflective tools.

ELIGIBILITY:
Inclusion Criteria:

* Persistent or recurrent pain lasting longer than 3 months
* Able to read and write English

Exclusion Criteria:

* Cancer (History of any bone-related cancer or cancer that metastasized to the bone; Currently in treatment for any cancer or plan to start cancer treatment in the next 12 months; History of any cancer treatment in the last 24 months)
* Active substance abuse
* Uncontrolled depression or psychosis
* Visual or hearing difficulties that would preclude participation
* Individuals started receiving disability or compensation within the past year, or currently involved in litigation
* Current/planned (in the next 2 years) enrollment in another study of a device or investigational drug that would interfere with this study, this may include participation in a blinded trial.
* Any other diseases or conditions that would make a patient unsuitable for study participation as determined by the site principal investigators. This would include but not be limited to severe psychiatric disorders, active suicidal ideations or history of suicide attempts, and an uncontrolled drug and/or alcohol addiction)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2023-04-25 (Actual); Primary Completion 2023-07-25 (Actual); Study Completion 2023-07-25 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Hannah Smotrich, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Reflective Process Group
Started | 23
Completed | 13
Not Completed | 10
Not completed — Principal Investigator Decision | 8
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Population: The difference between the number of participants at baseline and in the results was because of participant attrition and incomplete responses from participants that could not be included in the final results data.
Arm/Group | Reflective Process Group
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 18
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 4
  White | 16
  More than one race | 0
  Unknown or Not Reported | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 23

OUTCOME MEASURES:

1. Primary Outcome: Participants Engaged in the Interventions
Description: The timepoints were as follows: consent and survey (T1), Kick-off Meeting (T2), Workshop (T3), and Exit Interview (T4). Participants had to attend the Kick-off Meeting (T2) to be considered engaged in the intervention. Participants who did not attend the Kick-off Meeting (T2) were withdrawn. Participants who did not attend the Workshop (T3) could still attend the Exit Interview (T4).
Time Frame: Baseline (T1) to Exit Interview (T4), up to 68 days
Measure: Count of Participants; unit: Participants
Arm/Group | Reflective Process Group
Number analyzed (Participants) | 23
Participants
  Consent and Survey (T1) | 23
  Kick off Meeting (T2) | 14
  Workshop (T3) | 12
  Exit Interview | 13

2. Secondary Outcome: Patient Global Impression of Change (PGIC) at T4 Exit Interview
Description: Participants completed the PGIC at the exit interview. The PGIC had one question with seven options ranging from -3 to 3: very much worse (-3), much worse (-2), minimally worse (-1), no change (0), minimally improved (1), much improved (2), very much improved (3). A higher score indicated greater improvement since the start of the study.
Time Frame: at T4 Exit Interview, up to 68 days
Population: Results reflect the participants who attended the T4 exit interview and completed the PGIC. Of the 13 participants who attended the exit interview, 1 did not complete the PGIC.
Measure: Count of Participants; unit: Participants
Arm/Group | Reflective Process Group
Number analyzed (Participants) | 12
Participants
  Very much improved | 0
  Much Improved | 4
  Minimally Improved | 5
  No change | 2
  Minimally worse | 0
  Much worse | 1
  Very much worse | 0

3. Secondary Outcome: Change in Pain Interference Based on the Patient-Reported Outcomes Measurement Information System (PROMIS) 29 Version 2.0 Between Baseline (t1) and Approximately 68 Days (t4 Exit Interview)
Description: There were 4 questions in this questionnaire. For each question, participants selected one of five options, ranging from "not at all" (1) to "very much" (5). Total scores ranged from 4 to 20 points, where higher scores indicated more pain interference. Since this survey was discussing the change in the pain interference, a negative score indicated less pain interfering with day-to-day activities.The change betwen the baseline (T1 and Exit Interview (t4) is reported.
Time Frame: Up to 68 days
Population: The difference between the number of participants at baseline and in the results here is because of participant attrition and incomplete responses from participants that could not be included in the final results data.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Change in Reflective Process Group: Self-guided at home activities: After the kick-off meeting participants will complete the cultural probe kit for 3 weeks. This kit is a design research tool, to prompt participants to document, map, journal, and reflect on various aspects of daily lives. Following this, participants will attend a facilitated workshop and then complete the next at-home kits.
Arm/Group | Change in Reflective Process Group
Number analyzed (Participants) | 23
score on a scale
  Baseline | 13.833 (2.791)
  Change from Baseline to Exit Interview: number analyzed (Participants) | 12
  Change from Baseline to Exit Interview | -1.583 (3.753)

ADVERSE EVENTS:
Time Frame: Up to 45 days.
Description: Adverse event means any untoward medical occurrence, whether or not considered intervention-related (21 CFR 312.32 (a)). A serious adverse event is a death, life-threatening adverse event, inpatient or prolonged hospitalization, persistent or substantial disruption of normal life functions, or congenital anomaly/birth defect. Other important medical events may be considered serious if medical or surgical intervention is required to prevent one of the outcomes listed.
Arm/Group | Reflective Process Group
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-04-20): https://cdn.clinicaltrials.gov/large-docs/81/NCT05847881/Prot_SAP_001.pdf
  • Informed Consent Form (2023-04-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT05847881/ICF_000.pdf